CLINICAL TRIAL: NCT06538194
Title: Comparison of the Efficacy of Dextrose Prolotherapy and Mesotherapy in Lateral Epicondylitis: A Prospective Randomised Controlled Trial
Brief Title: Comparison of the Efficacy of Dextrose Prolotherapy and Mesotherapy in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sibel süzen Özbayrak, M.D., Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMU-GETAT-KAEK/27.03.2024/06
Record Dates: First submitted 2024-06-04; First posted 2024-08-05 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; mesotherapy; prolotherapy; elbow pain
MeSH Terms: conditions — Tennis Elbow | interventions — Mesotherapy; Prolotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mesotherapy (Active Comparator): The first group received mesotherapy: For this group, a solution containing 1 cc each of lidocaine, pentoxifylline, vitamin B complex diluted 1/10 with saline, thiocolchicoside, and meloxicam diluted 1/5 with saline will be made. A 30 gauge, 4 mm mesotherapy injector will be used for the application. The lateral epicondyle will be the site of an intradermal injection. Of that amount, 2.5 cc will be applied point-by-point at intervals of 1-2 cm, and the remaining 2.5 cc will be applied using the napage method, 0.1 cc of solution were given with each injection.
  Interventions: Procedure: Mesotherapy
- Prolotherapy (Active Comparator): Group 2 received dextrose prolotherapy: A 22 gauge syringe was used to apply a total of 5 cc of 15% dextrose solution (a combination of 3.75 ml 20% dextrose and 1.25 mg 2% lidocaine) to at least 5 most sensitive points of the lateral epicondyle. It was injected 3 times with 3 weeks intervals.
  Interventions: Procedure: Mesotherapy
- Control (Active Comparator): Only exercise and resting wrist splints will be administered to the third group, which is the control group.
  Interventions: Procedure: Mesotherapy

INTERVENTIONS:
Procedure: Mesotherapy — For 1. group, a solution containing 1 cc each of lidocaine, pentoxifylline, vitamin B complex diluted 1/10 with saline, thiocolchicoside, and meloxicam diluted 1/5 with saline will be made. A 30 gauge, 4 mm mesotherapy injector will be used for the application. The lateral epicondyle will be the site of an intradermal injection. Of that amount, 2.5 cc will be applied point-by-point at intervals of 1-2 cm, and the remaining 2.5 cc will be applied using the napage method, 0.1 cc of solution were given with each injection. This injection will be applied once a week for a total of 4 sessions. Group 2 received dextrose prolotherapy: A 22 gauge syringe was used to apply a total of 5 cc of 15% dextrose solution (a combination of 3.75 ml 20% dextrose and 1.25 mg 2% lidocaine) to at least 5 most sensitive points of the lateral epicondyle. It was injected 3 times with 3 weeks intervals.
  Other Names: Prolotherapy

SUMMARY:
A total of 84 patients with lateral epicondylitis were included in the study. The patients were randomly assigned to 3 treatment groups: mesotherapy (n = 28), prolotherapy (n = 28), and control (n = 28). Patients were evaluated before treatment and at the 3rd and 8th weeks of treatment for pain severity measured with the Visual Activity Scale (VAS) during resting, activity, and at night, and for functional status with a short version of the upper limb-specific disabilities of the arms, shoulder, and hand (Quick-Dash) and Oxford Elbow Score.

DETAILED DESCRIPTION:
This randomised-controlled single-blind prospective study was carried out at a Physical Medicine and Rehabilitation out-patient clinic. After approval by the Ethics Committee, all participants signed a written informed consent form. The research was conducted in accordance with the Helsinki Declaration.

Participants

The study will include individuals with lateral epicondylitis who are between the ages of 20 and 60 and have had elbow pain for at least three months. Pain around the lateral epicondyle during resisted extension of wrist and fingers and tenderness over the lateral epicondyle were required for the diagnosis of lateral epicondylitis. Patients with the following exclusion criteria were not accepted into the study:

* Recent upper-extremity surgery,
* Recent upper extremity trauma, fracture, or dislocation,
* Upper-extremity peripheral neuropathy,
* Infectious processes of joint or soft tissues of the upper extremity
* Decompensated heart or respiratory failure
* Rheumatologic Diseases
* Psychiatric Disorders
* History of allergy to ingredients of injection solution

Demographic informations were recorded. Severity of elbow pain in resting, activity and if present night pain were recorded according to Visual analogue Scale (VAS). Functional impairment were evaluated with short version of the upper limb-specific Disabilities of Arms, Shoulder and Hand (Quick-Dash) and Oxford Elbow Score.

Following clinical assessment, patients were divided into three treatment groups randomly. Mesotherapy, Prolotherapy and Control groups. Exercise and resting wrist splints were recommended for all groups.

The first group received mesotherapy: For this group, a solution containing 1 cc each of lidocaine, pentoxifylline, vitamin B complex diluted 1/10 with saline, thiocolchicoside, and meloxicam diluted 1/5 with saline will be made. A 30 gauge, 4 mm mesotherapy injector will be used for the application. The lateral epicondyle will be the site of an intradermal injection. Of that amount, 2.5 cc will be applied point-by-point at intervals of 1-2 cm, and the remaining 2.5 cc will be applied using the napage method, 0.1 cc of solution were given with each injection.

Group 2 received dextrose prolotherapy: A 22 gauge syringe was used to apply a total of 5 cc of 15% dextrose solution (a combination of 3.75 ml 20% dextrose and 1.25 mg 2% lidocaine) to at least 5 most sensitive points of the lateral epicondyle. It was injected 3 times with 3 weeks intervals.

Only exercise and resting wrist splints will be administered to the third group, which is the control group.

All measures were conducted at baseline, after treatment, at 3th and 8th weeks follow-ups.

ELIGIBILITY:
Inclusion Criteria:

Elbow pain for at least three months. Pain around the lateral epicondyle during resisted extension of wrist and fingers Tenderness over the lateral epicondyle

Exclusion Criteria:

* Recent upper-extremity surgery,
* Recent upper extremity trauma, fracture, or dislocation,
* Upper-extremity peripheral neuropathy,
* Infectious processes of joint or soft tissues of the upper extremity
* Decompensated heart or respiratory failure
* Rheumatologic Diseases
* Psychiatric Disorders
* History of allergy to ingredients of injection solution

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
VAS | All measures were conducted at baseline, after treatment, at 3th and 8th weeks follow-ups.
  Measurement of Pain Severity. The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10 cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
short version of the upper limb-specific Disabilities of Arms, Shoulder and Hand (Quick-Dash) | All measures were conducted at baseline, after treatment, at 3th and 8th weeks follow-ups.
  Measurement of Functional Disability. The possible score ranges from 0 to 100 points. 0 points represent a complete, unrestricted function of the upper extremities, while 100 points represent the greatest possible functional impairment. The DASH score is one of the most established questionnaires for disorders of the upper limb.
Oxford Elbow Score | All measures were conducted at baseline, after treatment, at 3th and 8th weeks follow-ups.
  Measurement of Functional Disability. The outcome can be interpreted based on a 48-point scale: 0-19, poor; 20-29, fair; 30-39, good; and 40-48, excellent

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Haydarpasa Numune Research and Training Hospital, Istanbul, Uskudar, Turkey (Türkiye)

REFERENCES:
- [Background] Arias-Vazquez PI, Castillo-Avila RG, Tovilla-Zarate CA, Quezada-Gonzalez HR, Arcila-Novelo R, Loeza-Magana P. Efficacy of prolotherapy in pain control and function improvement in individuals with lateral epicondylitis: A Systematic Review and Meta-analysis. ARP Rheumatol. 2022 Apr-Jun;1(2):152-167. PMID 35810374
- [Background] Piraccini E, Biondi G. Prolotherapy: Regenerative Medicine for Lateral Epicondylitis. Turk J Anaesthesiol Reanim. 2020 Dec;48(6):509-510. doi: 10.5152/TJAR.2020.82356. Epub 2020 May 18. PMID 33313593